Hip Fracture in Individuals under 60 Years of Age. A Prospective Multi-Center Study of the Epidemiology, Treatment, Outcome and Patient Satisfaction Regarding Hip Fractures.

Statistical analysis plan

10 February 2019

# 1.a. Bone quality, demographics and hormonal status in hip fracture patients under 60 years of age.

First author: Strøm Rönnquist

Co-authors: (in random order) Åkesson; Palm, Tange Kristensen, Bech Jensen; Fladmose

Madsen, Overgaard; Viberg.

Last author: Rogmark

Study design: Prospective multi-center cohort study *Participants*: Approx. 200 individuals aged 18-60 years

Exposure: Acute, non-pathological hip fracture (intra- and extracapsular), regardless of

trauma level

Control group: Cohorts of middle-aged, non-fractured individuals with DXA measurements

at Odense and Skåne University Hospital

Aim:

- 1. Comparison of bone mineral density at the time of hip fracture (DXA scan) and basic risk factors for osteoporosis (BMI, smoking, etc. = variables accessible in the control groups)

  Statistical analysis of categorical data using Chi-square test.
- 2. Descriptive analysis of other relevant factors in a young hip fracture cohort Statistical analysis of categorical data using Chi-square test.

Collected variables in the prospective study:

Gender, age, BMI

Comorbidity, medication

Diet

Abuse – alcohol, drugs, tobacco, anabolic steroids

Socioeconomics (working capacity, type of living)

Fracture history (own and first-hand relatives)

Laboratory tests including hormonal status

DXA scan at the time of the fracture

Fracture pattern, type of trauma

Physical / functional level prefracture (New mobility score and others)

Health-related quality-of-life prefracture

# Hypotheses:

There are differences in BMD and risk factors when comparing the hip fracture group with a standard control group.

Within the hip fracture group; different levels of BMD are associated with comorbidities, hormonal status and life style factors.

## Perspective/clinical relevance:

To identify those patients who have an underlying cause or reason for sustaining a hip fracture in relatively young age and, when appropriate, initiate preventive measures for future fractures.

# 1.b. Association between fracture type, fracture trauma type and bone mineral density

First author: Strøm Rönnquist

Co-authors: (in random order) Åkesson; Palm, Tange Kristensen; Fladmose Madsen,

Overgaard; Viberg. *Last author:* Rogmark

Study design: Prospective multi-center cohort study *Participants*: Approx. 200 individuals aged 18-60 years

Exposure: Acute, non-pathological hip fracture (intra- and extracapsular) regardless of trauma

level

Study groups: High and low bone mineral density; high and low trauma injuries.

Aim:

1. Analysis of association between bone mineral density at the time of hip fracture (DXA scan) and fracture type.

Statistical analysis of categorical data using Chi-square test.

2. Analysis of association between trauma type and fracture type.

Statistical analysis of categorical data using Chi-square test.

# Collected variables in the prospective study:

Fracture pattern (femoral neck fracture – undisplaced and displaced; basocervical fracture; trochanteric fracture – stable and unstable; subtrochanteric fracture)

Type of trauma (other than low-energy, low-energy)

DXA scan at the time of the fracture

For adjustment:

Gender, age, BMI

Comorbidity, medication

Diet

Abuse – alcohol, drugs, tobacco, anabolic steroids Socioeconomics (working capacity, type of living) Fracture history (own and first-hand relatives) Laboratory tests including hormonal status

Physical / functional level prefracture (New mobility score and others)

Health-related quality-of-life prefracture

#### Hypotheses:

There is no association between low BMD and displaced/unstable hip fracture

There is no association between higher trauma energy and displaced/unstable hip fracture.

There is an association when both low BMD and higher trauma energy exists and displaced/unstable hip fracture.

### Perspective/clinical relevance:

To understand the interaction between trauma energy level and bone strength (as measured by DXA) and fracture type.